CLINICAL TRIAL: NCT03228758
Title: Efficacy of Anterior Versus Posterior Myotomy Approach in Per Oral Endoscopic Myotomy (POEM) for the Treatment of Achalasia - A Single Operator Analysis
Brief Title: Anterior Orientation vs Posterior Orientation in Per Oral Endoscopic Myotomy POEM for the Treatment of Achalasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WUH 17008; 18-01666 (Other: NYULangone Institutional Review Board)
Record Dates: First submitted 2017-07-13; First posted 2017-07-25 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Achalasia
Keywords: POEM
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either the anterior or posterior orientation approach to the endoscopic myotomy.
Who Masked: Participant
Masking Description: Subjects will not be made aware of the orientation approach to the endoscopic myotomy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior Orientation (Active Comparator): The anterior endoscopic myotomy of the lower esophageal sphincter will be performed between the 11 o'clock to 3 o'clock position in the esophagus determined by the usual endoscopic convention of 12 o'clock representing the most anterior aspect of the esophagus on endoluminal view.
  Intervention is the endoscopic myotomy of the lower esophageal sphincter.
  Interventions: Procedure: Per Oral Endoscopic Myotomy
- Posterior Orientation (Active Comparator): The posterior endoscopic myotomy of the lower esophageal sphincter will be performed between the 5 o'clock to 6 o'clock position in the esophagus determined by the usual endoscopic convention of 12 o'clock representing the most anterior aspect of the esophagus on endoluminal view.
  Intervention is the endoscopic myotomy of the lower esophageal sphincter.
  Interventions: Procedure: Per Oral Endoscopic Myotomy

INTERVENTIONS:
Procedure: Per Oral Endoscopic Myotomy — The Per Oral Endoscopic Myotomy procedure is the cutting of the lower esophageal sphincter. This procedure is a natural orifice transluminal endoscopic surgery (NOTES)

SUMMARY:
The purpose of this study is to compare the safety and efficacy of the anterior versus posterior myotomy technique in Per Oral Endoscopic Myotomy (POEM) for the treatment of Achalasia. The primary efficacy outcome is periprocedural pain requiring the use of narcotics. The secondary outcomes focus on safety which includes technical procedure duration time; tunneling time, myotomy time, and closure time; incidence of mucosotomy (transmural and non-transmural injury), capnoperitoneum, and the postoperative sequelae of gastrointestinal reflux disease (GERD). Periprocedural pain data collection will include post POEM procedure pain scores, administrations of analgesia until discharge.

The final analysis will focus on determining whether there is a statistically significant difference in the amount and severity of pain in the Anterior versus Posterior myotomy subject populations. Additional analysis will be the collection of analgesic type (narcotic versus non-narcotic), dosage, frequency, and duration of treatment from post POEM procedure in the endoscopy recovery suite until the subjects are discharged.

DETAILED DESCRIPTION:
Achalasia is one of the most studied esophageal motility disorders. The etiology of Achalasia is autoimmune, neurodegenerative, or viral immune. Achalasia is a consequence of the degeneration of ganglion cells in the myenteric plexus of the esophageal body and the lower esophageal sphincter (LES). The end result of the inflammatory process is the loss of inhibitory neurotransmitters nitrous oxide and vasoactive intestinal peptide causing the imbalance between excitatory and inhibitory neurons. This results in failure of the lower esophageal sphincter (LES) to relax and is associated with aperistalsis of the esophageal body, leading to difficulty swallowing, food and fluid stasis; regurgitation of undigested food, fluid and saliva; and weight loss. Achalasia is an incurable disease and treatments are only focused on the relaxation of the lower esophageal sphincter in order to allow for passage of food fluid and saliva into the stomach. It has an estimated prevalence of 10 cases per 100,000 populations and an incidence of 1-3 cases per 100,000 populations per year in the Western world.

The armamentarium of Achalasia treatment includes pharmacologic management with the use of calcium channel blockers, nitrites, phosphodiesterase inhibitor (sildenafil), anticholinergics, and beta-adrenergic agonists; endoscopy using botulinum toxin injections just above the squamocolumnar junction or pneumatic balloon dilation of the lower esophageal sphincter; open Heller Myotomy, laparoscopic Heller Myotomy, and Per Oral Endoscopic myotomy (POEM). Per oral endoscopic myotomy (POEM) is the most recent innovative treatment in the armamentarium of Achalasia treatment. Per oral endoscopic myotomy (POEM) is a natural orifice transluminal endoscopic surgery (NOTES) approach to a Heller myotomy for the treatment of Achalasia. In 2008, POEM was first performed successfully in a human subject by Haruhiro Inoue in Japan. The POEM was performed on a 36 year old patient without any documented post-operative complications. In 2009, Stavros Stavropoulos at Winthrop University Hospital (WUH) performed the first per oral endoscopic myotomy (POEM) procedure outside of Japan. The POEM was performed on a 42 year old male without documented post-operative complications. The subject had a marked improvement in objective manometric and barium esophagram findings; and improvement in subjective dysphagia score. Consequently there has been a rapidly increasing volume of POEM procedures performed in Japan, China, and throughout the United States. Stavropoulos at Winthrop University Hospital has the highest single-operator volume in the United States. The performance of POEM is still in evolution with various centers around the world performing variations on technique.

The International Per Oral Endoscopic Myotomy Survey (IPOEMS) was conducted by Stavropoulos and Savides during the July 2012 annual meeting of Natural Orifice Surgery Consortium for Assessment and Research (NOSCAR). This survey was conducted to address the scarceness of POEM literature at the time. IPOEM provided a "snapshot" of the status of POEM worldwide. The survey included 5 Asian, 7 North American, and 4 European expert centers with a combined total of 841 POEM procedures performed by July 2012. At the time most centers (14) performed right anterior myotomy (2 o'clock orientation) with only a few of centers performing posterolateral myotomy (5 o'clock orientation) determined using the usual endoscopic convention of 12 o'clock representing the most anterior aspect of the esophagus on endoluminal view.

The esophagus in humans is a complex structure with multiple muscles, nerves, vascular, and lymphatic components. Branches of the vagus nerve and visceral branches of the sympathetic trunk provide nerve fibers to the esophageal plexus. The vagus nerve delivers two fiber types to the esophageal plexus: preganglionic parasympathetic fibers and afferent fibers. These vagal fibers in the esophageal plexus reform to make the anterior vagal trunk (left vagus) and the posterior vagal trunk (right vagus). The anterior and posterior terms for the vagal trunks are used in relation to the esophagus. The visceral branches of the sympathetic trunk delivers two fiber types to the esophageal plexus: sympathetic postganglionic fibers and the afferent fibers. The afferent fibers originating from the sympathetic trunk are primarily involved with pain. The critical anatomical component of the esophagus in the treatment of Achalasia is the lower esophageal sphincter. Per common convention, the most anterior point of the LES point is assigned as the 12 o'clock position. The strong oblique sling fiber component is centered at 7o'clock on the posterolateral wall and wraps over the anterior and posterior walls at 11 o'clock and 5 o'clock, respectively. The weaker circular clasp fiber component location is centered at 2 o'clock to 3 o'clock. The question of investigating the optimal orientation to perform the myotomy is unique to POEM. Open Heller myotomy and laparoscopic Heller myotomy are limited to the anterior aspect of the esophagus. Myotomy orientation is constrained by the anatomical locations of the left bronchus, left atrium and spine. Anterior orientation is forced between the 1 o'clock - 2 o'clock position secondary to the locations of the left bronchus and left atrium between 10 o'clock -11 o'clock and 12 o'clock - 1 o'clock, respectively. Posterior orientation is forced between the 4 o'clock - 5 o'clock positions secondary to the location of the spine located between 8 o'clock-9 o'clock positions .The sling fibers maintain the angle of His and are a significant antireflux barrier. Stavropoulos et al, reported on a single operator series of 284 POEM subjects at Digestive Disease Week in May 2016. A statistical difference was found in the number of subjects requiring narcotics post POEM procedure Subjects who had an anterior myotomy were less likely to require narcotics post POEM procedure than those subjects who had a posterior myotomy, 35% versus 53% respectively (p=0.007).

To date, there have been no prospective randomized controlled studies conducted comparing anterior versus posterior myotomy technique in POEM analyzing perioperative pain, procedure duration, incidence of mucosotomy, capnoperitoneum, and the postoperative sequelae of gastrointestinal reflux disease (GERD).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have been diagnosed with Achalasia Type I, II, or III by positive manometric findings and supporting findings by timed barium esophagram and endoscopy.
2. Subjects who are willing and competent to sign Informed Consent and to comply with study related visits and procedures.

Exclusion Criteria:

1. Subjects who are under 18 years of age
2. Subjects with Achalasia Type I, II, or III who have had a prior failed open or laparoscopic Heller myotomy; or have an esophageal diverticula, or anatomical variant dictating the approach of the myotomy
3. Subjects diagnosed with other motility disorders such as distal esophageal spasm (DES), hypertensive peristalsis (Nutcracker), or hypercontractile esophagus (Jackhammer)
4. Subjects with coagulopathy
5. Pregnant females
6. Subjects who in the investigators' opinion, are medically unstable , are unable to give informed consent, or whose risks outweigh the benefits of participating in the study
7. Subjects with decisional incapacity who are unable to comply with study related visits and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2019-05-24 (Actual)

PRIMARY OUTCOMES:
Periprocedural pain requiring the use of narcotics. | Within the first 48 hours after the procedure.
  Pain related to the endoscopic myotomy requiring the use of narcotic pain medication.

SECONDARY OUTCOMES:
Incidence of Gastrointestinal Reflux Disease (GERD) | Within 3 months after the procedure.
  Gastrointestinal Reflux Disease measured by BRAVO pH study

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Stavropoulos, MD, Principal Investigator — NYU Langone Winthrop
Locations (1):
- NYU Winthrop Hospital, Mineola, New York, United States

REFERENCES:
- [Result] Nguyen NQ, Holloway RH. Recent developments in esophageal motor disorders. Curr Opin Gastroenterol. 2005 Jul;21(4):478-84. PMID 15930992
- [Result] Vaezi MF, Pandolfino JE, Vela MF. ACG clinical guideline: diagnosis and management of achalasia. Am J Gastroenterol. 2013 Aug;108(8):1238-49; quiz 1250. doi: 10.1038/ajg.2013.196. Epub 2013 Jul 23. PMID 23877351
- [Result] Walzer N, Hirano I. Achalasia. Gastroenterol Clin North Am. 2008 Dec;37(4):807-25, viii. doi: 10.1016/j.gtc.2008.09.002. PMID 19028319
- [Result] Ruffato A, Mattioli S, Lugaresi ML, D'Ovidio F, Antonacci F, Di Simone MP. Long-term results after Heller-Dor operation for oesophageal achalasia. Eur J Cardiothorac Surg. 2006 Jun;29(6):914-9. doi: 10.1016/j.ejcts.2006.03.044. Epub 2006 May 3. PMID 16675239
- [Result] Ujiki MB, Yetasook AK, Zapf M, Linn JG, Carbray JM, Denham W. Peroral endoscopic myotomy: A short-term comparison with the standard laparoscopic approach. Surgery. 2013 Oct;154(4):893-7; discussion 897-900. doi: 10.1016/j.surg.2013.04.042. PMID 24074429
- [Result] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Result] Richter JE. Update on the management of achalasia: balloons, surgery and drugs. Expert Rev Gastroenterol Hepatol. 2008 Jun;2(3):435-45. doi: 10.1586/17474124.2.3.435. PMID 19072391
- [Result] Stavropoulos SN, Harris MD, Hida S, Brathwaite C, Demetriou C, Grendell J. Endoscopic submucosal myotomy for the treatment of achalasia (with video). Gastrointest Endosc. 2010 Dec;72(6):1309-11. doi: 10.1016/j.gie.2010.04.016. No abstract available. PMID 21111876
- [Result] Stavropoulos SN, Modayil RJ, Friedel D, Savides T. The International Per Oral Endoscopic Myotomy Survey (IPOEMS): a snapshot of the global POEM experience. Surg Endosc. 2013 Sep;27(9):3322-38. doi: 10.1007/s00464-013-2913-8. Epub 2013 Apr 3. PMID 23549760
- [Result] Stavropoulos, SN, Modayil, R, and Brathwaite, et al. Anterior vs. posterior per oral endoscopic myotomy (POEM): Is there a difference in outcome? Gastrointest Endosc 2016; 83 (5S): AB145
- [Result] Friedel D, Modayil R, Stavropoulos SN. Per Oral Endoscopic Myotomy (POEM): review of current techniques and outcomes (including postoperative reflux). Curr Surg Rep 2013; 1: 203-213.
- [Result] Stranding, S. (2016) Mediastinum, In Gray's anatomy: the anatomical basis of clinical practice. (41st Ed.). (pp. 976-993) Elsevier Limited in Clinical Key Flex